CLINICAL TRIAL: NCT03460769
Title: Evaluation of a Mixed Meal Test for Diagnosis and Characterization and Type 3c Diabetes Mellitus Secondary to Pancreatic Cancer and Chronic Pancreatitis (DETECT)
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0742 (PA17-0674); 1U01DK108328-01 (NIH); NCI-2018-02275 (Other: NCI-Clinical Trials Registry)
Record Dates: First submitted 2018-02-07; First posted 2018-03-09 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer; Chronic Pancreatitis; Diabetes Mellitus Type 3c
Keywords: Pancreatic Cancer; Chronic Pancreatitis; Diabetes Mellitus Type 3c; Data management
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sample collection (CP and PDAC groups): During the mixed meal tests, blood samples will be collected at a fasting baseline (time 0 min), then 15, and 30 minutes following meal ingestion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pancreatic Cancer: The Coordinating and Data Management Center (CDMC) at MD Anderson Cancer will be responsible for the coordination and data management for the Evaluation of a mixed meal test for Diagnosis and characterization of Type 3c diabetes mellitus secondary to pancreatic cancer and chronic pancreatitis (DETECT).
  Interventions: Other: Data Management and Monitoring
- Chronic Pancreatitis: The Coordinating and Data Management Center (CDMC) at MD Anderson Cancer will be responsible for the coordination and data management for the Evaluation of a mixed meal test for Diagnosis and characterization of Type 3c diabetes mellitus secondary to pancreatic cancer and chronic pancreatitis (DETECT).
  Interventions: Other: Data Management and Monitoring
- Type 3c Diabetes Mellitus: The Coordinating and Data Management Center (CDMC) at MD Anderson Cancer will be responsible for the coordination and data management for the Evaluation of a mixed meal test for Diagnosis and characterization of Type 3c diabetes mellitus secondary to pancreatic cancer and chronic pancreatitis (DETECT).
  Interventions: Other: Data Management and Monitoring

INTERVENTIONS:
Other: Data Management and Monitoring — The Coordinating and Data Management Center (CDMC) at MD Anderson Cancer responsible for the coordination and data management for the Evaluation of a mixed meal test for Diagnosis and characterization of Type 3c diabetes mellitus secondary to pancreatic cancer and chronic pancreatitis (DETECT), which is part of the NIH U01 funded Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer (CPDPC).

SUMMARY:
The Coordinating and Data Management Center (CDMC) at MD Anderson Cancer will be responsible for the coordination and data management for the Evaluation of a mixed meal test for Diagnosis and characterization of Type 3c diabetes mellitus secondary to pancreatic cancer and chronic pancreatitis (DETECT), which is part of the NIH U01 funded Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer (CPDPC). Similar to all studies that will be coordinated and managed by the CDMC, no patient enrollment will occur at MDACC. All patient recruitment will occur at external sites that are a part of the CPDPC, which are listed in the appended DETECT protocol. The data management systems, auditing, and monitoring effort are supported by the CDMC.

DETAILED DESCRIPTION:
Objectives:

1. Evaluate the pancreatic polypeptide response following a standardized mixed meal in new onset diabetes associated with PDAC (particularly with a proximal tumor) and chronic pancreatitis vs. T2DM.
2. Evaluate the insulin and glucagon response following a standardized mixed meal in new onset diabetes associated with PDAC and chronic pancreatitis vs. T2DM.
3. Evaluate the incretin response following a standardized mixed meal in new onset diabetes associated with PDAC and chronic pancreatitis vs. T2DM.
4. Explore the differences in analytes from Objectives 1-3 in a cohort of subjects with the same diseases and long-standing DM or normoglycemia.
5. Evaluate differences in fasting levels of insulin and novel biomarkers in pancreatic cancer compared to chronic pancreatitis and T2DM.
6. Explore the metabolic alterations (including pancreatic polypeptide response and insulin secretion) in diabetes associated with pancreatic surgery for chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* All Participants must sign an informed consent indicating that they are aware of the investigational nature of this study. Participants must have signed an authorization for the release of their protected health information.
* Participants must be ages ≥30 and <85.
* Participants must have a diagnosis of one of the following based on study definitions;
* New Onset Diabetes (<3 years) in participants with Pancreatic Cancer (PDAC);
* New Onset Diabetes (<3 years) in participants with Chronic Pancreatitis;
* New Onset Diabetes (<3 years) in participants without Pancreatic disease (i.e., T2DM)
* Long standing T2DM (≥3 years) without Pancreatic disease
* Long standing diabetes (≥3 years) in participants with PDAC
* Long standing diabetes (≥3 years) participants with chronic pancreatitis
* non-diabetic participants with PDAC
* non-diabetic participants with chronic pancreatitis
* non-diabetic controls without Pancreatic disease

Exclusion Criteria:

* Participants must not have any significant medical illnesses (including diabetes) that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the Participant's ability to tolerate study interventions.
* Diabetes not stable enough to permit holding of diabetes medications in Participants undergoing mixed meal tolerance testing.
* Participants taking higher doses of insulin (≥0.75 unit/kg/day). [Criterion is not applicable for PDAC Participants undergoing fasting only blood collection]
* Participants in the non-pancreatic disease subgroup on longer acting agents, including thiazolidinediones and once-weekly GLP-1 agonists (Bydureon [exenatide], Ozempic [semaglutide], Trulicity [dulaglutide]). [Criterion is not applicable for Participants in the CP and PDAC groups].
* Participants currently receiving oral steroid medications.
* Hospitalization for acute pancreatitis within 2 months before study visit. [Criterion is not applicable for PDAC Participants undergoing fasting only blood collection]
* The presence of a symptomatic cyst in Participants with CP. [Criterion is not applicable for PDAC Participants undergoing fasting only blood collection; this includes cancer arising from a mucinous cystic lesion].
* Any Participant with a known pancreatic cancer histologic subtype other than adenocarcinoma (e.g., Participants with pancreatic neuroendocrine tumors are excluded).
* Previous pancreatic surgery (including total pancreatectomy, pancreaticoduodenectomy, distal pancreatectomy, pancreaticojejunostomy, enucleation, or Frey procedure). [Criterion is not applicable for CP Participants with diabetes who have a history of pancreaticoduodenectomy, pancreaticojejunostomy, distal pancreatectomy, or Frey].
* Previous treatment for pancreatic cancer, including chemotherapy or radiation.
* Previous vagotomy or gastric surgery, including endoscopic gastric reduction procedures. [Criterion is not applicable for PDAC Participants undergoing fasting only blood collection].
* Previous diagnosis of gastroparesis. [Criterion is not applicable for PDAC Participants undergoing fasting only blood collection].
* Participants on treatment for any cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix).
* Allergy or intolerance to ingredients in Boost drink in Participants undergoing mixed meal testing (see Appendix 13.9) [Criterion is not applicable for PDAC Participants undergoing fasting only blood collection].

Ages: 30 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants recruited from external sites.
Sampling Method: Non-Probability Sample
Enrollment: 775 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Protocol and Regulatory Compliance Monitoring of Regulatory Documents for Consortium Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer (CPDPC) | 3 years
  The Coordinating and Data Management Center (CDMC) at MD Anderson Cancer Center will monitor protocol and regulatory compliance at all participating institutions.

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Chari, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (10):
- United States (10):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Florida, Gainesville, Florida
  - Indiana University, Carmel, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Hart PA, Kudva YC, Yadav D, Andersen DK, Li Y, Toledo FGS, Wang F, Bellin MD, Bradley D, Brand RE, Cusi K, Fisher W, Mather K, Park WG, Saeed Z, Considine RV, Graham SC, Rinaudo JA, Serrano J, Goodarzi MO. A Reduced Pancreatic Polypeptide Response is Associated With New-onset Pancreatogenic Diabetes Versus Type 2 Diabetes. J Clin Endocrinol Metab. 2023 Apr 13;108(5):e120-e128. doi: 10.1210/clinem/dgac670. PMID 36404274
- See also: MD Anderson Cancer Center — http://www.mdanderson.org